CLINICAL TRIAL: NCT01045590
Title: Phase IV, Multicenter, Single-blind, Positive-controlled, Parallel Group Study of Glibenclamide (Dose to be Titrated From Starting Dose of 5mg om) Plus Rosiglitazone 4mg om (Increased to 8mg om After 6 Months) and vs Glibenclamide (Dose to be Titrated With Starting Dose of 5mg om) Plus Placebo, Adm
Brief Title: Glibenclamide (Dose to be Titrated From Starting Dose of 5mg om) Plus Rosiglitazone 4mg om (Increased to 8mg om After 6 Months) and vs Glibenclamide (Dose to be Titrated With Starting Dose of 5mg om) Plus Placebo, Administered to Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 100684
Record Dates: First submitted 2009-12-10; First posted 2010-01-11 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2011-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- glibenclamide + Rosiglitazone (Active Comparator): glibenclamide plus rosiglitazone
  Interventions: Drug: titration
- glibenclamide + placebo (Placebo Comparator)
  Interventions: Drug: titration

INTERVENTIONS:
Drug: titration — Patients in the glibenclamide plus placebo treatment group Patients in the glibenclamide plus placebo treatment group who have FPG < 270mg/dL after the glibenclamide 5mg om run-in will continue to receive glibenclamide 5mg om. At every subsequent visit, the glibenclamide dose will be titrated to achieve the target HbA1c level of < 7%. If the HbA1c is > 7%, the dose of glibenclamide will be escalated in the following sequence: from 5mg om, to 5mg om, 2.5mg on, to 5mg bd and 7.5mg om, 5mg on, to 7.5mg bd. The maximum total daily dose will not exceed 15 mg. A downward titration of glibenclamide using the above sequence in the reverse order can be used to maintain normoglycemia at any visit. Once the target HbA1c level of < 7% is achieved, the dose of glibenclamide is maintained. If at the glibenclamide dose of 7.5mg bd, the HbA1c is > 7% for 2 subsequent visits, the patient will be withdrawn from the study.
  Arms: glibenclamide + placebo
Drug: titration — Patients in the glibenclamide + rosiglitazone treatment group who have FPG < 270mg/dL after the glibenclamide 5mg om run-in will receive glibenclamide 5mg om + rosiglitazone 4mg om. At every subsequent visit, the glibenclamide dose will be titrated to achieve the target HbA1c level of < 7%. If the HbA1c is > 7%, the dose of glibenclamide will be escalated in a similar fashion as above. The only exception is at visit 5 when the dose of rosiglitazone is increased (see next paragraph). Once the target HbA1c level of < 7% is achieved, the dose of glibenclamide is maintained. If at the glibenclamide dose of 7.5mg bd, the HbA1c is > 7% for 2 subsequent visits, the patient will be withdrawn from the study.
  Arms: glibenclamide + Rosiglitazone

SUMMARY:
Rationale Rosiglitazone and troglitazone both promote differentiation of pre-adipocytes into adipocytes in subcutaneous, but not omental fat, and reduce gamma glutamyl transferase, a surrogate marker for intra-abdominal and hepatic fat. Troglitazone has been shown by abdominal computed tomography (CT) and magnetic resonance imaging (MRI) scan to reduce the intra-abdominal adipose tissue area in type 2 diabetics. Similarly rosiglitazone has also been shown to increase subcutaneous but not intra-abdominal fat in patients with type 2 diabetes. In the same study it was also shown to cause a substantial reduction in hepatic fat. Central fat depots are believed to be associated with more cardiovascular risk than subcutaneous fat depots. By contrast, sulphonylurea-associated weight gain has been shown by abdominal CT scan to include increases in intra-abdominal adipose tissue.

The aim of this study is to compare the body fat distribution pattern of glibenclamide plus rosiglitazone versus glibenclamide and placebo (especially the intra-abdominal adipose tissue and abdominal subcutaneous adipose tissue areas) in patients with type 2 diabetes. It is hypothesised that rosiglitazone will lead to the accumulation of excess energy stores in the subcutaneous rather than the intra-abdominal adipose tissue depot. In addition, it is hoped that by having a positive effect on diastolic blood pressure, lipid levels, BMI, rosiglitazone will be shown to have a better cardiovascular risk profile when used in combination with glibenclamide rather than when glibenclamide is used alone.

Although insulin resistance has been shown to be a primary defect causing type 2 diabetes mellitus, insulin secretory defect has also been known to be an important factor in the development of type 2 diabetes mellitus. A previous study has shown that in Korean patients, early-phase insulin secretory defect may be the initial abnormality in the development of type 2 diabetes mellitus [56].

This study also aims to assess the efficacy and safety of glibenclamide plus rosiglitazone versus glibenclamide plus placebo therapy in Korean patients with type 2 diabetes. In addition, a previous study has shown that in Korean patients, early-phase insulin secretory defect may be the initial abnormality in the development of type 2 diabetes mellitus. This study aims to show that rosiglitazone treatment in Korean patients, regardless of their early phase insulin secretory ability, is just as efficacious and safe.

Objective(s) Primary To evaluate the effect of 12 months oral treatment with glibenclamide plus rosiglitazone versus oral glibenclamide plus placebo, on body fat distribution (as measured by the change in the ratio between the intra-abdominal adipose tissue and abdominal subcutaneous adipose tissue areas) in patients with type 2 diabetes.

Secondary

* To investigate the efficacy of glibenclamide plus rosiglitazone, compared to glibenclamide plus placebo on beta-cell function and insulin resistance as calculated by HOMA-B and HOMA-R.
* To investigate the efficacy of glibenclamide plus rosiglitazone, compared to glibenclamide plus placebo on fasting plasma glucose, insulin, fasting serum lipid profile (total cholesterol, triglycerides, HDL cholesterol, LDL cholesterol and total cholesterol to HDL cholesterol ratio).
* To investigate the efficacy of glibenclamide plus rosiglitazone, compared to glibenclamide plus placebo on early phase insulin secretion during an oral glucose tolerance test as measured by the insulinogenic index.
* To define further the clinical safety and tolerability of glibenclamide plus rosiglitazone through the assessment of physical examinations, vital signs, weight, routine laboratory tests, adverse experiences and electrocardiograms (ECGs).

Endpoint(s) Primary Change from baseline in the ratio (IAAT:SAT) between the intra-abdominal adipose tissue area (IAAT) and abdominal subcutaneous adipose tissue area [SAT] after 12 months treatment with oral glibenclamide plus rosiglitazone compared to oral glibenclamide plus placebo Secondary

Comparisons will be made between glibenclamide plus rosiglitazone and glibenclamide plus placebo treatment groups on Change from baseline after 6 and 12 months treatment with respect the following:

CT Scan

Derived from CT image at the lumbar IV level:

* abdominal subcutaneous adipose tissue area [SAT]
* intra-abdominal adipose tissue area [IAAT]

Derived from the CT image of the right leg at the thigh level (1cm below the gluteal fold):

* total subcutaneous adipose tissue area [TSAT] Derived from CT images at the lumbar IV and thigh level
* ratio between abdominal subcutaneous adipose tissue area [SAT] and total subcutaneous adipose tissue area of the thigh [TSAT]
* ratio between intra-abdominal adipose tissue area [IAAT] and total subcutaneous adipose tissue area of the thigh [TSAT] Derived from Oral Glucose Tolerance Test, glycaemic response to OGTT, difference

ELIGIBILITY:
Subjects were selected by following considerations:

* Diagnosis of type 2 diabetes mellitus defined by the American Diabetic Association (ADA) criteria.
* Subject whose diabetes was managed by diet, exercise, and/or sulfonylurea, and/or metformin, who could be converted to treatment with glibenclamide 5mg om.
* 126mg/dL ≤ fasting plasma glucose (FPG) ≤ 270mg/dL and HbA1c level >7% at screening. In addition, the following criterion was applied prior to randomization: 126mg/dL ≤ fasting plasma glucose (FPG) ≤ 270mg/dL at baseline(after 2 months of run-in treatment with glibenclamide 5mg om only).

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-12; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the ratio (IAAT:SAT) between the intra-abdominal adipose tissue area (IAAT) and abdominal subcutaneous adipose tissue area [SAT] after 12 months treatment with oral glibenclamide plus rosiglitazone compared to oral glibenclamide p | baseline

SECONDARY OUTCOMES:
Comparisons will be made between glibenclamide plus rosiglitazone and glibenclamide plus placebo treatment groups on Change from baseline after 6 and 12 months treatment with respect the following | baseline

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Seoul, South Korea